CLINICAL TRIAL: NCT04780360
Title: Evaluation of Post Operative Pain, Early Wound Healing, and the Time of Application of Cyanoacrylates Tissue Adhesives Versus Silk Sutures at the Palatal Donor Area of Subepithelial Connective Tissue Grafts (CTG) A Randomized Clinical Trial: Comparative Study
Brief Title: Cyanoacrylate Tissue Adhesives Versus Silk Suture at the Palatal Donor Site of Sub Epithelial Connective Tissue Graft
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed Saeed Mohamed Ibrahuim Abdullah, Researcher, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 567
Record Dates: First submitted 2019-11-17; First posted 2021-03-03 (Actual); Last update posted 2021-03-08 (Actual); Status verified 2021-03

CONDITIONS: The Effect of Local Aplication of Cayanoacrylate Tissue Adhesives on Improving the Healing

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cayanoacrylate tissue adhesives (Experimental): thin layers of high viscosity blend of n-butyl and 2-octyl cayanoacrylate tissue adhesive will be applied and rinsed with saline at least three times with interval of at least 30 seconds
  Interventions: Procedure: Cayanoacrylate tissue adhesives
- Silk suture material (Active Comparator): interrupted knots
  Interventions: Procedure: Silk suture

INTERVENTIONS:
Procedure: Cayanoacrylate tissue adhesives — Cyanoacrylates are a family of strong fast-acting adhesives with industrial, medical, and household uses. They are various esters of cyanoacrylic acid. The acryl groups in the resin rapidly polymerize in the presence of water to form long, strong chains
  Arms: Cayanoacrylate tissue adhesives
Procedure: Silk suture — Non Absorbalble suture materiel used to fixed the edges of the incision in place until healing
  Arms: Silk suture material

SUMMARY:
Subepithelial connective tissue grafts (CTG) are considered the gold standard procedure with proven clinical success when it comes to gingival augmentation aims to to improve periodontal health, which can enhance the long-term prognosis of teeth by obtaining soft tissue coverage of exposed root surfaces and/or augmentation the dimensions of gingival tissue. The procedure require harvesting tissue from a the palate, which increases the complexity of the procedure and patient discomfort. Complications after harvesting a graft would be pain, inflammation, bleeding, flap necrosis and infection in the donor site.

ELIGIBILITY:
Inclusion Criteria:

* Patients with mucogingival defects scheduled for sub epithelial connective tissue graft
* Age at least 18 years.
* Not having any systemic disease that could compromise wound healing
* No periodontal surgery on the experimental sites.
* No smoking,
* No pregnancy or lactation

Exclusion Criteria:

* Patients with coagulation disorders
* patients on corticosteroids, with uncontrolled diabetes, or with any systemic disease that precluded periodontal surgery
* patients with a history of contact dermatitis to formaldehyde
* Loss of maxillary premolars and molars
* Medications or antibiotics used in the previous 6 months
* Pregnancy or lactation
* Smoking

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-12-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Early Wound Healing | 1 week
  Measured By Modified Early Wound Healing Index

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Cairo Universty, Cairo, Egypt